CLINICAL TRIAL: NCT00478972
Title: A Randomized, Double-blind, Placebo-controlled, Parallel-group, Fixed Single-dose Regimen, Multicenter Study to Assess the Efficacy and Safety of SR141716 in Obese Type 2 Diabetic Patients Inadequately Controlled With Diet and Exercise Alone
Brief Title: Japanese Study With Rimonabant in Obese Type 2 Diabetic Patients on Diet and Exercise
Acronym: SOLO
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Company decision taken in light of demands by certain national health authorities
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EFC6648
Record Dates: First submitted 2007-05-24; First posted 2007-05-25 (Estimated); Last update posted 2016-06-08 (Estimated); Status verified 2016-06

CONDITIONS: Obesity; Diabetes Mellitus Type 2
Keywords: obese; diabetes; cannabinoid-1 receptor
MeSH Terms: conditions — Obesity; Diabetes Mellitus, Type 2; Diabetes Mellitus | interventions — Rimonabant; Diet; Exercise

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Rimonabant (Experimental): Rimonabant 20 mg once daily in addition to diet and exercise
  Interventions: Drug: Rimonabant; Other: Diet and exercise
- Placebo (Placebo Comparator): Placebo (for Rimonabant) once daily in addition to diet and exercise
  Interventions: Drug: placebo (for Rimonabant); Other: Diet and exercise

INTERVENTIONS:
Drug: Rimonabant — Tablet, oral administration
  Other Names: SR141716; Acomplia
  Arms: Rimonabant
Drug: placebo (for Rimonabant) — Tablet, oral administration
  Arms: Placebo
Other: Diet and exercise — Target daily caloric intake: Ideal body weight × 25 kcal

SUMMARY:
The primary objective of this study is to assess the efficacy of Rimonabant (SR141716) compared to placebo on change in HbA1c and on relative change in body weight over 36 weeks in obese type 2 diabetic patients inadequately controlled with diet and exercise alone.

The secondary objectives are:

* To evaluate the effect of Rimonabant compared to placebo on other parameters related to the glucose control, waist circumference, Body Mass Index and metabolic parameters;
* To evaluate the safety and tolerability of Rimonabant compared to placebo;
* To evaluate the pharmacokinetics of Rimonabant.

DETAILED DESCRIPTION:
The total duration per patient will be approximately 53 weeks including a 36-week double-blind treatment period.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 Diabetes Mellitus patients inadequately treated with diet and exercise alone (not drug treated)
* HbA1C ≥ 7.0 % and ≤ 10.0 %
* Body Mass Index ≥ 25 kg/m²

Exclusion Criteria:

* Type 1 diabetes
* Within 12 weeks prior to screening visit: use of oral antidiabetic drugs and/or insulin, of anti-obesity drugs or other drugs for weight reduction
* Within 4 weeks prior to screening visit: administration of systemic long-acting corticosteroids or prolonged use (more than one week) of other systemic corticosteroids, change in lipid lowering treatment
* Secondary obesity
* Primary hyperlipidemia
* Positive serum pregnancy test in females of childbearing potential

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 321 (Actual)
Dates: Start 2007-04; Primary Completion 2009-01 (Actual); Study Completion 2009-01 (Actual)

PRIMARY OUTCOMES:
Absolute change from baseline in HbA1C | Baseline to Week 36
Relative change from baseline in body weight | Baseline to Week 36

SECONDARY OUTCOMES:
Absolute change from baseline in Fasting Plasma Glucose | Baseline to Week 36
Absolute change from baseline in waist circumference | Baseline to Week 36
Relative change from baseline in Triglycerides and HDL-cholesterol | Baseline to Week 36
Safety: Overview of adverse events | Baseline to Week 47

CONTACTS AND LOCATIONS:
Overall Officials: ICD CSD, Study Director — Sanofi
Locations (1):
- Sanofi-Aventis Administrative Office, Tokyo, Japan